CLINICAL TRIAL: NCT05296005
Title: Total Neoadjuvant Therapy for the Treatment of Gastroesophageal Junction (GEJ) and Gastric Cancers: A Pilot Trial
Brief Title: Neoadjuvant Therapy for the Treatment of Gastroesophageal Junction and Gastric Cancers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20191; NCI-2021-11289 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-13; First posted 2022-03-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage IIA Gastric Cancer AJCC v8; Clinical Stage IIB Gastric Cancer AJCC v8; Clinical Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Gastric Adenocarcinoma; Pathologic Stage IB Gastric Cancer AJCC v8; Pathologic Stage IC Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage II Gastric Cancer AJCC v8; Pathologic Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIA Gastric Cancer AJCC v8; Pathologic Stage IIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIB Gastric Cancer AJCC v8; Pathologic Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8
MeSH Terms: interventions — Capecitabine; Docetaxel; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; Radiotherapy; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, chemoradiation, surgery) (Experimental): NEOADJUVANT CHEMOTHERAPY: Patients receive FLOT chemotherapy consisting of docetaxel intravenously (IV) , oxaliplatin IV, leucovorin IV, and fluorouracil IV over 24 hours on day 1 or FOLFOX chemotherapy consisting of oxaliplatin IV and leucovorin IV, and fluorouracil IV continuously over 24 hours on days 1 and 2. Treatment repeats every 2 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.
  NEOADJUVANT CHEMORADIATION: Within 4 weeks after completing neoadjuvant chemotherapy, patients undergo radiation therapy in 25 fractions over 5 weeks. Patients also receive either fluorouracil IV continuously for 24 hours on days 1-5 or capecitabine orally (PO) twice daily (BID) on days 1-5. Cycles repeat weekly for 5 weeks in the absence of disease progression or unacceptable toxicity.
  SURGERY: Within 4-8 weeks after neoadjuvant chemoradiation, patients undergo surgical resection according to tumor location and per surgeon expertise.
  Interventions: Drug: Capecitabine; Drug: Docetaxel; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Radiation: Radiation Therapy; Procedure: Surgical Procedure

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Radiation: Radiation Therapy — Undergo radiotherapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Surgical Procedure — Undergo surgical resection
  Other Names: Operation; Surgery; Surgery Type; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase I trial tests the safety, side effects studies chemotherapy followed by chemotherapy at the same time as radiation therapy (chemoradiation) before surgery (neoadjuvant) in treating patients with stage gastric (stomach) or gastroesophageal junction cancer . Chemotherapy drugs, such as docetaxel, oxaliplatin , leucovorin, fluorouracil, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving chemotherapy and chemoradiation before surgery may make the tumor smaller and may reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of delivering tailored targeted neoadjuvant therapy with chemotherapy followed by chemoradiation and surgery in patients with gastroesophageal junction gastroesophageal junction (GEJ) and gastric cancer.

II. To assess the toxicity of delivering tailored targeted neoadjuvant therapy with chemotherapy followed by chemoradiation and surgery in patients with GEJ and gastric cancer.

SECONDARY OBJECTIVES:

I. To identify the resident microbiota species associated with higher response to the combination therapy and quantify abundance and diversity of favorable bacterial communities over the course of the therapy.

II. To evaluate local control, progression-free survival, and overall survival at 3, 6, 9, 12 and 24 months after treatment with neoadjuvant chemotherapy and chemoradiation.

III. To describe the perfusion and early tumor uptake kinetics of primary tumor targets at baseline, during and following systemic chemotherapy and chemoradiation therapies using 18F-fluorodeoxyglucose (18F-FDG) digital photon counting positron emission tomography/computed tomography (dPET/CT) approaches.

IV. To evaluate 18F-FDG dPET/CT to evaluate and characterize residual primary tumor following neoadjuvant chemotherapy and initial chemoradiation therapy for subsequent adaptive boost radiation delivery.

EXPLORATORY OBJECTIVE :

I. To explore FDG dPET standardized uptake value (SUV) metrics (e.g., SUVmax, SUVpeak, SUVmax Tumor-to-Liver, SUVpeak Tumor-to-Liver, metabolic tumor volume, etc.) on early dynamic PET perfusion, early tumor FDG uptake and delayed tumor FDG uptake to better predict pathologic response of primary tumor following multimodality therapy and surgical resection.

OUTLINE:

NEOADJUVANT CHEMOTHERAPY: Patients receive FLOT chemotherapy consisting of docetaxel intravenously (IV) , oxaliplatin IV, leucovorin IV, and fluorouracil IV over 24 hours on day 1 or FOLFOX chemotherapy consisting of oxaliplatin IV and leucovorin IV, and fluorouracil IV continuously over 24 hours on days 1 and 2. Treatment repeats every 2 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity.

NEOADJUVANT CHEMORADIATION: Within 4 weeks after completing neoadjuvant chemotherapy, patients undergo radiation therapy in 25 fractions over 5 weeks. Patients also receive either fluorouracil IV continuously for 24 hours on days 1-5 or capecitabine orally (PO) twice daily (BID) on days 1-5. Cycles repeat weekly for 5 weeks in the absence of disease progression or unacceptable toxicity.

SURGERY: Within 4-8 weeks after neoadjuvant chemoradiation, patients undergo surgical resection according to tumor location and per surgeon expertise.

After completion of study treatment, patients are followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven, cT2N0-T4aN3M0 (TNM 8th edition), gastric or Siewert II-III GEJ adenocarcinoma
* Evaluation with endoscopic ultrasound (EUS) and staging laparoscopy prior to enrollment is strongly recommended.
* Patient should be a candidate for neoadjuvant chemotherapy with fluorouracil, leucovorin, oxaliplatin and docetaxel (FLOT) or fluorouracil and oxaliplatin (FOLFOX).
* Patients should be >= 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patient should be eligible for surgical intervention
* T1 N0 disease (assessed by endoscopic ultrasound)

Exclusion Criteria:

* Evidence of distant metastatic disease
* Solitary functioning kidney within the potential radiation field
* Peripheral polyneuropathy > National Cancer Institute (NCI) grade II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients able to complete all planned procedures and interventions successfully | Up to 24 months
Incidence of adverse events | Up to within 30 days of discontinuation of protocol treatment

SECONDARY OUTCOMES:
Resident microbiota species associated with higher response | Up to 24 months
Time to progression | From date of treatment completion to the event of interest or otherwise censored at last follow-up, assessed up to 12 months
Progression-free survival (PFS) | From date of treatment completion to the event of interest or otherwise censored at last follow-up, assessed up to 12 months
  Kaplan-Meier analysis will be used to estimate PFS. PFS will include any failure (local, regional, or distant) or death from any cause.
Overall survival (OS) | From date of treatment completion to the event of interest or otherwise censored at last follow-up, assessed up to 12 months
  Kaplan-Meier analysis will be used to estimate OS. OS will be death from any cause.
Perfusion and early tumor uptake kinetics of primary tumor using 8F-FDG dPET/CT approaches | Up to 25 months
  To describe the perfusion and early tumor uptake kinetics of primary tumor targets at baseline, during and following systemic chemotherapy and chemoradiation therapies using 18F-FDG dPET/CT approaches
18F-FDG dPET/CT to evaluate and characterize residual primary tumor following neoadjuvant chemotherapy and initial chemoradiation therapy for subsequent adaptive boost radiation delivery. | Up to 12 months

OTHER OUTCOMES:
Standard uptake value SUVmax metrics | Up to 24 months
  Will explore 18F-fluorodeoxyglucose (FDG) digital photon counting positron emission tomography (dPET) SUV metrics (e.g., SUVmax, SUVpeak, SUVmax Tumor-to-Liver, SUVpeak Tumor-to-Liver, metabolic tumor volume, etc.) on early dynamic PET perfusion, early tumor FDG uptake and delayed tumor FDG uptake to better predict pathologic response of primary tumor following multimodality therapy and surgical resection.
Standard uptake value SUVpeak Tumor-to-liver metrics | Up to 24 months
  Will explore 18F-fluorodeoxyglucose (FDG) digital photon counting positron emission tomography (dPET) SUV metrics (e.g., SUVmax, SUVpeak, SUVmax Tumor-to-Liver, SUVpeak Tumor-to-Liver, metabolic tumor volume, etc.) on early dynamic PET perfusion, early tumor FDG uptake and delayed tumor FDG uptake to better predict pathologic response of primary tumor following multimodality therapy and surgical resection.
Standard uptake value metabolic tumor volume metrics | Up to 24 months
  Will explore 18F-fluorodeoxyglucose (FDG) digital photon counting positron emission tomography (dPET) SUV metrics (e.g., SUVmax, SUVpeak, SUVmax Tumor-to-Liver, SUVpeak Tumor-to-Liver, metabolic tumor volume, etc.) on early dynamic PET perfusion, early tumor FDG uptake and delayed tumor FDG uptake to better predict pathologic response of primary tumor following multimodality therapy and surgical resection.
Standard uptake value SUVmax Tumor-to-liver metrics | Up to 24 months
  Will explore 18F-fluorodeoxyglucose (FDG) digital photon counting positron emission tomography (dPET) SUV metrics (e.g., SUVmax, SUVpeak, SUVmax Tumor-to-Liver, SUVpeak Tumor-to-Liver, metabolic tumor volume, etc.) on early dynamic PET perfusion, early tumor FDG uptake and delayed tumor FDG uptake to better predict pathologic response of primary tumor following multimodality therapy and surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Dayssy A Diaz Pardo, MD, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu